CLINICAL TRIAL: NCT02098798
Title: Comparison of Surveillance Colonoscopy Techniques in Patients With IBD
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Iacucci Marietta MD,PhD, Clinical Associate Professor, University of Calgary
Other Study IDs: REB13-0960
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Inflammatory Bowel Disease
Keywords: Dysplasia, Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HD: High Definition Colonoscopy alone
  Interventions: Procedure: HD Colonoscopy
- HD + iSCAN: HD colonoscopy + iSCAN
  Interventions: Procedure: HD Colonoscopy + iSCAN
- HD + Dye: High definition colonoscopy + dye spraying chromoendoscopy
  Interventions: Procedure: HD Colonoscopy + dye spray

INTERVENTIONS:
Procedure: HD Colonoscopy — High definition colonoscopy procedure in surveillance colonoscopy
  Groups: HD
Procedure: HD Colonoscopy + iSCAN
  Groups: HD + iSCAN
Procedure: HD Colonoscopy + dye spray
  Groups: HD + Dye

SUMMARY:
We propose a randomized controlled study to determine the detection rates of neoplasia with high definition colonoscopy alone, high definition dye spraying chromoendoscopy or High definition iSCAN virtual chromoendoscopy in patients with long standing colitis (8 years from diagnosis except primary sclerosing cholangitis when surveillance starts at diagnosis) CD or UC.

We hypothesized that these novel endoscopic techniques using High definition colonoscopy with virtual chromoendoscopy -iScan 2 and 3 may be superior to high definition colonoscopy alone and similar to using dye spraying chromoendoscopy for detection of dysplasia and neoplasia in patients with long standing IBD.

We will aim to demonstrate if we can avoid dye spraying during the procedure and save expense and considerable time.

In addition, we can hope to produce evidence and inform the way in which we perform surveillance colonoscopy especially without large number of multiple random biopsies but only few targeted" smart and intelligent" biopsies using high definition colonoscopy with iSCAN technique as is already the European practice in several centres.

ELIGIBILITY:
Inclusion Criteria:

Clinical and histological diagnosis of UC or colonic CD-extensive or pancolitis.

UC -CD Disease duration 8 years from diagnosis UC-CD with associated primary sclerosing cholangitis from diagnosis Ulcerative Colitis Activity Index Mayo score 0-1 (inactive disease) Crohn's disease Activity Index - Harvey Bradshaw score <4 (dysplasia detection requires quiescent inflammatory bowel disease)

Exclusion Criteria:

Known intraepithelial neoplasia or colorectal cancer or other neoplasia Coagulopathy which may prevent biopsies Pregnancy Inability to obtain informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inflammatory bowel disease patients undergoing surveillance colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Detection of neoplasia in the 3 cohorts - high definition colonoscopy, HD colonoscopy + iSCAN, HD colonoscopy + dye chromoendoscopy | At the time of procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Foothills Medical Centre, Calgary, Alberta, Canada